CLINICAL TRIAL: NCT05658146
Title: An Open-label, Randomized, Single-dose, Three-way Crossover Study to Establish Bioequivalence of 5 mg Mavacamten Capsule 1 and 5 × 1 mg Mavacamten Capsule 2 to 5 mg Mavacamten Capsule 2 in Healthy Participants
Brief Title: A Study to Assess the Effects on the Single-Dose Drug Levels of Mavacamten in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV027-1052
Record Dates: First submitted 2022-12-13; First posted 2022-12-20 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; Mavacamten; Bioequivalence
MeSH Terms: interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental)
  Interventions: Drug: Mavacamten Capsule 1; Drug: Mavacamten Capsule 2; Drug: Mavacamten Capsule 3
- Sequence 2 (Experimental)
  Interventions: Drug: Mavacamten Capsule 1; Drug: Mavacamten Capsule 2; Drug: Mavacamten Capsule 3
- Sequence 3 (Experimental)
  Interventions: Drug: Mavacamten Capsule 1; Drug: Mavacamten Capsule 2; Drug: Mavacamten Capsule 3
- Sequence 4 (Experimental)
  Interventions: Drug: Mavacamten Capsule 1; Drug: Mavacamten Capsule 2; Drug: Mavacamten Capsule 3
- Sequence 5 (Experimental)
  Interventions: Drug: Mavacamten Capsule 1; Drug: Mavacamten Capsule 2; Drug: Mavacamten Capsule 3
- Sequence 6 (Experimental)
  Interventions: Drug: Mavacamten Capsule 1; Drug: Mavacamten Capsule 2; Drug: Mavacamten Capsule 3

INTERVENTIONS:
Drug: Mavacamten Capsule 1 — Specified dose on specified days
  Other Names: BMS-986427, MYK-461
Drug: Mavacamten Capsule 2 — Specified dose on specified days
  Other Names: BMS-986427, MYK-461
Drug: Mavacamten Capsule 3 — Specified dose on specified days
  Other Names: BMS-986427, MYK-461

SUMMARY:
The purpose of this study is to assess the effects on the single-dose drug levels of mavacamten in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 32 kilograms/meter squared (kg/m^2) inclusive, at the screening visit.
* Healthy, as determined by physical examination, vital signs, electrocardiograms (ECGs), and clinical laboratory assessments (including hematology, chemistry, and urinalysis) within the normal range at the screening visit and/or on Day -1.
* Cytochrome P450 (CYP) 2C19 normal, rapid, or ultrarapid metabolizer, as determined by genotyping during screening.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Current or history of clinically significant cardiac condition, including but not limited to arrhythmia, left ventricular systolic dysfunction, coronary heart disease; current, history, or family history of hypertrophic cardiomyopathy; or evidence of prior myocardial infarction based on ECGs.
* CYP2C19 poor (*2/*2, *3/*3, or *2/*3) or intermediate (*1/*2, *1/*3, *2/*17) metabolizer, as determined by genotyping during screening.
* Use of CYP2C19 and CYP3A4 inducers or inhibitors within 28 days of study intervention administration.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | From Day 1 up to Day 35±2 of each period
Area Under the Serum Concentration-time Curve from Time Zero to Time of Last Quantifiable Concentration [AUC(0-T)] | From Day 1 up to Day 35±2 of each period
Area Under the Serum Concentration-time Curve from Time Zero Extrapolated to Infinite Time [AUC(INF)] | From Day 1 up to Day 35±2 of each period

SECONDARY OUTCOMES:
Area Under the Serum Concentration-time Curve from Time 0 to 72 Hours [AUC(0-72)] | From Day 1 to Day 4 of each period
Time of Maximum Observed Serum Concentration (Tmax) | From Day 1 up to Day 35±2 of each period
Terminal Half-life (T-HALF) | From Day 1 up to Day 35±2 of each period
Number of Participants with Adverse Events (AEs) | Up to 35 days post discontinuation of dosing
Number of Participants with Serious Adverse Events (SAEs) | Up to 35 days post discontinuation of dosing
Number of Participants with Vital Sign Abnormalities | Up to 35 days post discontinuation of dosing
Number of Participants with Electrocardiograms (ECG) Abnormalities | Up to 35 days post discontinuation of dosing
Number of Participants with Physical Examination Abnormalities | Up to 35 days post discontinuation of dosing
Number of Participants with Clinical Laboratory Evaluation Abnormalities | Up to 35 days post discontinuation of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution - 0001, Anaheim, California
  - Local Institution - 0002, Miami, Florida
  - Local Institution - 0003, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html